CLINICAL TRIAL: NCT07342309
Title: Real-World Treatment Patterns and Outcomes of Patients With HER2-Altered Metastatic Breast Cancer in the United States
Brief Title: Real-World Treatment Patterns and Outcomes in HER2-Altered Metastatic Breast Cancer Patients in the United States
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1479-0045
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Metastatic breast cancer cohort (mBC): Adult patients (>=18 years) with confirmed diagnosis of recurrent or de novo metastatic breast cancer (mBC) who were diagnosed between January 1, 2018, through March 31, 2024 (1 year prior to the data cutoff date, March 31, 2025) in the Flatiron Solid Tumor Discovery Clinico-Genomic Database (CGDB).
- HER2-positive subcohort (mBC HER2+): Patients meeting eligibility of the mBC cohort.
  Evidence of HER2 positive (HER2+) as defined by immunohistochemistry (IHC)/in situ hybridization (ISH)
  * IHC 3+ or
  * IHC 2+ and evidence of HER2 amplification by ISH or
  * ISH+ without further information on IHC.
- HER2-mutant subcohort (mBC HER2-mutant): Patients meeting eligibility of the mBC cohort.
  Evidence of NGS short variant alterations at any time in the database, regardless of the functional type, which includes missense, nonsense, frameshift, nonframeshift, or splice variants.
  Patients who are not included in the HER2+ subcohort.

SUMMARY:
This study aims to address the following key objectives in patients with HER2-altered mBC:

Primary objectives

* Estimate the prevalence of human epidermal growth factor receptor 2 positive (HER2+), human epidermal growth factor receptor 2 (HER2) mutation, cooccurrence of HER2+ and HER2 mutation among adult patients with metastatic breast cancer (mBC)
* Among mBC patients with HER2+ and HER2 mutation, describe the following:

  * Baseline demographic and clinical characteristics
  * Treatment patterns during follow-up including 1L through fifth-line (5L) settings
  * Real-world overall survival (rwOS) for 1L through 5L

Secondary objectives

- Among mBC patients with HER2+ and HER2 mutation, examine the following (as permissible in the study data):

* Real-world progression-free survival (rwPFS)
* Real-world time to discontinuation (rwTTD)
* Real-world time to next treatment (rwTTNT)
* Real-world overall response rate (rwORR)

ELIGIBILITY:
Inclusion criteria:

Overall metastatic breast cancer (mBC) cohort (total population):

* Histologically or cytologically confirmed diagnosis of breast cancer (BC)
* Patient has at least 2 documented clinical visits in the Flatiron network, on different days, during the study period from 1 January 2011 through 31 March 2025
* Initial diagnosis of de novo or recurrent mBC established during the case selection window from 1 January 2018 through 31 March 2024 (1 year prior to the data cutoff date, 31 March 2025)

  -- The date of initial mBC diagnosis will define the study index date
* Aged ≥ 18 years at the study index date

Human epidermal growth factor receptor 2 (HER2)-positive subcohort (mBC HER2+):

* Patients meeting eligibility for the mBC cohort
* Patients can be HER2-mutant or HER2 nonmutant
* Evidence of HER2+ as defined by immunohistochemistry (IHC)/in situ hybridization (ISH) based on a test performed within 180 days before or 180 days after the index date. If a patient does not have any IHC/ISH test during the 180-day periods before or after the index date, then tests performed at any time in the pre-index date period will be examined and any evidence of HER2+ status will classify the patient as HER2+.

  * IHC 3+ or IHC 2+ and evidence of HER2 amplification by ISH or ISH+ (without further information on IHC) according to American Society of Clinical Oncology/College of American Pathologists guidelines.
  * The sample date will be used to define biomarker status. If the sample date is missing, the report date will be used.

HER2-mutant subcohort (mBC HER2-mutant):

* Patients meeting eligibility for the mBC cohort
* HER2-mutant: Patients are classified as having an HER2 mutation if there is evidence of NGS short variant alterations at any time in the database, regardless of the functional type, which includes missense, nonsense, frameshift, nonframeshift, or splice variants.

Exclusion criteria

mBC cohort (total population):

-To ensure adequate treatment and outcome data, any patient without a visit or medication record (i.e., medication order/administration or LOT) within 90 days of mBC diagnosis (i.e., the time window from 90 days before to 90 days after the mBC diagnosis).

HER2+ subcohort (mBC HER2+):

- None (other than those applicable for the mBC cohort).

HER2-mutant subcohort (mBC HER2-mutant):

- Patients who are included in the HER2+ subcohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>=18 years) with confirmed diagnosis of recurrent or de novo metastatic breast cancer (mBC) who were diagnosed between January 1, 2018, through March 31, 2024 (1 year prior to the data cutoff date, March 31, 2025) in the Flatiron Solid Tumor Discovery Clinico-Genomic Database (CGDB).
Sampling Method: Non-Probability Sample
Enrollment: 7933 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Real-world overall survival (rwOS) | Up to 15 years
  OS as an event for each patient will be defined as the date of death minus the index date + 1. For patients with no record of death, OS will be censored at the last visit date, defined as the date of the last visit of any type prior to data cutoff.
  Month and year of death are noted in the Flatiron Discovery Clinico-Genomic Database (CGDB); the day of death will be imputed as the midpoint (15 th) of the month of death.
  Endpoint will be assessed separately from the study index date (mBC diagnosis) and each of the line of therapy (LOT) index dates.

SECONDARY OUTCOMES:
Real-world time to treatment discontinuation (rwTTD) | Up to 15 years
  rwTTD is defined as the time from the LOT start date to the end of the LOT + 1 (inclusive of maintenance therapies associated with the main therapeutic regimen).
  End of LOT will be defined as a composite of discontinuation (with or without subsequent LOT) or death.
  Patients on treatment at the end of the study period will be censored at that date.
Real-world time to next treatment (rwTTNT) | Up to 15 years
  rwTTNT is defined as the difference between subsequent LOT index dates (e.g., time from the 1L start date to the 2L start date, time from 2L start date to the 3L start date).
  Patients not receiving a subsequent treatment line will be censored at the last visit date.
Real-world overall response rate (rwORR) | Up to 15 years
  rwORR will be computed as the proportion of patients who achieved either a complete response or a partial response at any time during the therapy line. Distribution of best responses will be reported only for patients with known clinical responses (excluding unknown and missing/not available) for each treatment line.
  Endpoint will be assessed separately for each LOT.
Real-world progression-free survival (rwPFS) | Up to 15 years
  rwPFS will be defined as the difference between the index date and first record of disease progression or death after the index date + 1.
  For patients with no record of disease progression, rwPFS will be censored at the start of a subsequent LOT or the date of the last clinical note before the end of the study period, whichever is earlier.
  Endpoint will be assessed separately from each of the LOT index dates.

CONTACTS AND LOCATIONS:
Locations (1):
- Ridgefield, Ridgefield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore, limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com